CLINICAL TRIAL: NCT03614052
Title: Efectividad de la Tamsulosina Como Tratamiento Adyuvante Previo a Ureterolitotomia Endoscopica
Brief Title: Tamsulosin as Adjuvant Treatment Prior to Endoscopic Ureterolithotomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems with the number of participants
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 171229002
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Ureterolithiasis; Ureteral Calculi; Urolithiasis
MeSH Terms: conditions — Ureterolithiasis; Ureteral Calculi; Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tamsulosin hydrochloride (Experimental): Tamsulosin hydrochloride 0,4 mg tablets by mouth per day for 5 days before ureteroscopy
  Interventions: Drug: Tamsulosin Hydrochloride 0.4 milligrams
- Placebo oral tablet (Placebo Comparator): Placebo oral tablets by mouth per day for 5 days before ureteroscopy
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride 0.4 milligrams — Tamsulosin hydrochloride 0,4mg for 5 days before ureteroscopic treatment of urolithiasis
  Other Names: tamsulosin0,4mg
  Arms: tamsulosin hydrochloride
Drug: Placebo Oral Tablet — Placebo oral tablet 1 tablet per day for 5 days before ureteroscopic treatment of urolithiasis
  Other Names: placebo
  Arms: Placebo oral tablet

SUMMARY:
This a study aiming to compare treatment with tamsulosin versus placebo in patients undergoing endoscopic treatment for urolithiasis. The main outcome is the rate of stone free patients.

DETAILED DESCRIPTION:
Endoscopic treatment of urolithiasis has increased during the last several years. Adrenergic receptors have been described mainly in the distal ureter. Blockage of adrenergic receptors has been associated to a decrease in ureteral resistance. In this study the investigators hypothesized that alpha blockers are associated to a decrease in ureteral resistance with an increase in successful endoscopic management of urolithiasis.

Only patients with urolithiasis undergoing to endoscopic treatment are offered to participate. Patients are randomized between placebo arm or tamsulosin 0.4 mg/day. Demographic characteristics, stones characteristics and information related to surgery are recorded. Main study outcome is stone free rate and successful insertion of semirigid ureteroscope 8,0 - 9,8 Fr. All patients are follow-up for 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urolithiasis undergoing to endoscopic ureterolithotomy

Exclusion Criteria:

* Patients with previous ureteral catheter

  * Patients with allergy to tamsulosin
  * Patients currently in treatment with tamsulosin for other disease different than ureterolithiasis
  * Multiple ureterolithiasis
  * Patients with impairment of their mental status

    * Patients with open surgeries in the affected ureter or urinary diversion
    * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
stone free rate | 30 days
  stone free rate after ureteroscopic management of urolithiasis

SECONDARY OUTCOMES:
failed ureteroscopy rate | 05 days
  failed ureteroscopy insertion in patient with urolithiasis secondary to a non accommodating ureter

CONTACTS AND LOCATIONS:
Overall Officials: Gaston Astroza, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico Pontificia Universidad católica de Chile, Santiago, Santiago Metropolitan, Chile